CLINICAL TRIAL: NCT05928533
Title: Performance Of Cervical Restorations Using Nitric Acid and Mineral Enriched Adhesive Versus Phosphoric Acid and Universal Adhesive: Randomized Clinical Trial.
Brief Title: Performance Of Cervical Restorations Using Nitric Acid and Mineral Enriched Adhesive Versus Phosphoric Acid and Universal Adhesive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourane Yasser Ali Mohamed Yassin, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nourane Yasser Ali Mohamed
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Clinical Performance
Keywords: clinical performance, cervical caries, bioactive restoration, nitric acid, universal adhesive
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scotchbond Etchant gel ,Single Bond Universal adhesive , Filtek Supreme flowable composite of 3M (Active Comparator): After cavity preparation, enamel and dentin will be etched for 15 seconds using Scotchbond Universal Etchant gel 3M. The surface will be rinsed for 10 seconds and dried with compressed air, removing all excess moisture without desiccating the dentin structure then apply two coats of Single Bond Universal adhesive 3M with a micro brush with rubbing action for 20 seconds then evaporate the solvent with gentle air stream until no movement is noticed in the adhesive then finally light cured for 10 seconds. A Filtek Supreme 3M flowable composite will be used to restore the prepared cavity after selecting the appropriate shade. The shade selection for the flowable composite will be done before the cavity preparation. The flowable composite will be applied in increments of 2mm thickness then light cured for 40 seconds using LED light curing unit.
- clean and boost enamel cleanser, RE GEN universal adhesive & flowable composite of vista apex. (Experimental): After cavity preparation, clean and boost enamel cleanser of vista apex will be used to clean enamel and dentin surface by three steps: 1. With the enclosed flow-thru brush tip, apply Clean & Boost to the surface to be cleansed, ensuring the surface is completely saturated. 2. Using the delivery brush tip, agitate the Clean & Boost on the surface for 10 seconds. 3. Rinse thoroughly. The RE GEN universal adhesive from vista apex will be applied with micro brush with rubbing action then air agitation. RE GEN Bio active flowable composite form vista apex will be added to the universal adhesive and then cured together for 20 seconds according to the manufacture instructions.

INTERVENTIONS:
Other: clean and boost enamel cleanser of vista apex , RE GEN universal adhesive from vista apex , RE GEN Bio active flowable composite form vista apex — the clean and boost use to clean the tooth surface after cavity preparation without causing severe form of hypersensitivity then the RE GEN universal adhesive is applied by using a brush and cured with the RE GEN flowable composite for 20 seconds. Curing both together increase the bioactivity of the material.

SUMMARY:
To evaluate the clinical performance of multifunction Nitric acid etch, mineral enriched adhesive and flowable resin composite liner versus the universal adhesive in etch and rinse mode and regular flowable liner in cervical carious anterior cavities.

DETAILED DESCRIPTION:
The annual failure of composite restoration represents 1 to 5 % with anterior teeth and 1 to3 % with posterior teeth . Many challenges appeared to be the causative factors of this failure such as the technique sensitivity of its placement, polymerization shrinkage, type and design of the cavity, location of the tooth, adhesive materials used last but not least operator and patient related factors. Some of these obstacles can be controllable and others cannot. According to the systematic review published in 2022, the most common reasons for composite failure are marginal deterioration which led consequently to secondary caries, marginal discoloration and post operative sensitivity. Restoration of the cervical carious lesions represents a great challenge to the restorative dentist due to the complicated clinical situation which include difficult isolation, variation in the tooth substrates and intraoral biomechanical challenges. Lots of modifications in the resin composite material and technique of application have been done and they are still ongoing to overcome the abovementioned inherited shortcomings.

The smear layer is considered as an unstable structure that affects the chemical and mechanical bonding between the restoration and tooth structure. There are different techniques to deal with the smear layer, either to remove, modify or dissolve it. Total removal of this layer with35-37% Phosphoric was the most used technique for preparing the tooth substrate to receive resin composite restoration. However, postoperative sensitivity was a repeated complaint from the patients. Selective enamel etching technique was introduced to solve this problem by only applying the phosphoric acid on the enamel margins and the multimode adhesive incorporating mild acidic monomer will achieve the dentin conditioning mission. Later, it was concluded that the clinical performance of multimode adhesives with etch, and rinse mode was better than with self-etch mode. Furthermore, there is available commercial product introduced to deal with the tooth substrate in a different way which is the multifunction nitric acid etch. It contains acid which enable the etching ability and cauterize the minor bleeding, isopropyl alcohol which acts as an antibacterial agent and cleans the surface before bonding and Hydroxyethyl methacrylate (HEMA) is a desensitizer which block the dentinal tubules to reduce the hypersensitivity.

Another concern, which can maximize the performance of the restorative system is the implementation of the bioactive property in the restorative system. The concept of bioactivity was achieved by introducing materials which interact with the surrounding tissues and produce a specific effect in the form of biological response or release of active substances. This release encourages remineralization and improves health, longevity and tissue regeneration. The idea of bioactivity was first introduced in dentistry by Larry Hench in 1960. Furthermore, the bioactive materials have many properties like inhibition of the bacterial growth by releasing calcium, sodium, silica and phosphate ion and an osteogenic property due to the use of calcium phosphate or tricalcium phosphate . Many trials were conducted to study the influence of using the bioactive materials in the restorative dentistry as the addition of fluoride, calcium phosphate particles and bioactive glass. The first used bioactive glass in dentistry was 45S5 glass in 1988. It is considered as a rich source of minerals which plays an important role in tooth remineralization. The remineralization is considered nowadays the most effective way to compensate the loss in tooth structure . Giomer is considered one of the most common categories of the bioactive materials. It relies on the incorporation of the surface pre reacted glass ionomer particles in its composition. Another category is termed as mineral enriched restorative system which incorporates bioactive glass in its composition . Such bio constructive materials work in conjugation with the healing ability of the human body to help in reinforcement of the tooth substrate. The bioactive glass is calcium sodium phosphosilicate based material which releases calcium and phosphate, increases the pH and optimizing the conditions for remineralization. Also, it contains hydrated silica which aids in the formation of hydroxyapatite like layers on the surface of restoration preventing the penetration of bacteria and secondary caries development. By adding the bioactive material, the restorative system will be able to survive for an extended time. Unfortunately, reviewing the literature revealed absence of any clinical trials that study the performance of multifunction nitric acid etch and the mineral enriched adhesive and flowable resin composite.

ELIGIBILITY:
Inclusion Criteria:

* Cervical carious anterior lesions.
* Age: (18-45Ys)
* Gender: male and female
* Low and moderate caries risk patient

Exclusion Criteria:

* Patients with poor oral hygiene.
* Presence of para functional habits.
* Systemic diseases or severe medical complications.
* Lack of compliance.
* Rampant caries.
* Xerostomia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Post operative sensitivity | 24hours, 6, 12 and18 months
  Modified USPHS criteria United states public health service

SECONDARY OUTCOMES:
Marginal deterioration | 24 hours,6,12 and 18 months
  Modified USPHS criteria United states public health service
Marginal discoloration | 24 hours, 6, 12 and 18 months
  Modified USPHS criteria United states public health service
Retention | 24 hours,6,12 and 18 months
  Modified USPHS criteria United states public health service
Secondary caries | 24 hours,6,12 and 18 months
  Modified USPHS criteria United states public health service

CONTACTS AND LOCATIONS:
Overall Officials: Olfat El sayed Hassanein, Professor, Study Director — Olfat.hassanein@dentistry.cu.edu.eg
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: June 2023- January 2025
Access Criteria: Norane yasser (Principle investigator), through a folder saved on the computer with password